CLINICAL TRIAL: NCT02711722
Title: Reduced Unloading in NAVA Improves Distribution of Ventilation in ICU Patients
Brief Title: NAVA Unloading - Effects on Distribution of Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peter Sackey, Associate professor, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/521-31/4
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Acute Respiratory Failure
Keywords: Neurally adjusted ventilatory assist
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PScli1 (Active Comparator): Patients are ventilated in Pressure support (PS) according to the Clinical settings for 30min.
  Interventions: Device: PScli1
- NAVAcli (Active Comparator): Patients are ventilated in Neurally Adjusted Ventilatory Assist (NAVA) and the assist is set in order to match to respiratory muscle unloading reached with PScli1. Patients are ventilated in NAVAcli for 30min.
  Interventions: Device: Neurally adjusted ventilatory assist
- NAVA40% (Active Comparator): Patients are ventilated in Neurally Adjusted Ventilatory Assist (NAVA) and the assist is set in order to target 40% muscle unloading based on the Neuro-Ventilatory Efficiency (NVE) measurement. Patients are ventilated in NAVA40% for 30min.
  Interventions: Device: Neurally adjusted ventilatory assist
- NAVA60% (Active Comparator): Patients are ventilated in Neurally Adjusted Ventilatory Assist (NAVA) and the assist is set in order to target 60% muscle unloading based on the Neuro-Ventilatory Efficiency (NVE) measurement. Patients are ventilated in NAVA60% for 30min.
  Interventions: Device: Neurally adjusted ventilatory assist
- PScli2 (Active Comparator): Patients return to PS ventilation, according to the Clinical settings as in PScli1 for 30min.
  Interventions: Device: PScli2

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist — Ventilation supported by NAVA
  * Blood gas analysis
  * Respiratory Parameters At the end of the study step Neuro-Ventilatory Efficiency and Neuro-Mechanical Efficiency are measured.
  Other Names: NAVA
  Arms: NAVA40%; NAVA60%; NAVAcli
Device: PScli1 — Pressure support set by clinicians prior to inclusion
  Other Names: Pressure support
  Arms: PScli1
Device: PScli2 — Pressure support at the same level as prior to the study
  Other Names: Pressure support
  Arms: PScli2

SUMMARY:
Title: Reduced Unloading in NAVA Improves distribution of Ventilation in ICU patients.

Objectives:

1. To investigate if NAVA targeted to moderate respiratory muscular unloading results in redistribution of ventilation to the dorsal regions of the lungs
2. To verify if the redistribution of ventilation translates to a better gas exchange and to a potentially lung protective ventilation strategy (lower airway pressures)
3. To verify the possibility to set NAVA at different levels of unloading, based on Neuro-Ventilatory Efficiency.

Study Design: Randomised Crossover of Pressure Support and NAVA at different levels of unloading.

Population: Adult Intubated patients at the Neurosurgical ICU, ventilated for more than 48h, in weaning phase from mechanical ventilation.

Study duration: 2,5h Number of subjects: 12

DETAILED DESCRIPTION:
Critically ill patients on mechanical ventilation are at risk for developing respiratory muscle atrophy. Partial Assist modes such Pressure Support (PS) and Neurally Adjusted Ventilatory Assist (NAVA) are developed to maintain patients´own effort in breathing. However there are no recommendations on how to set the optimal ventilator support in NAVA to avoid over- or underassistance.

A previous Electrical Impedance Thomography (EIT) study has shown a redistribution of ventilation towards the dorsal regions of the lung in acute lung injury patients ventilated with NAVA, compared to PS.

In the present study, the assist is targeted to different respiratory muscle unloading, predefined and based on the Neuro-Ventilatory Efficiency (NVE). The NVE will be measured at 10min intervals and NAVA level adjusted if needed, to keep constant the level of unloading in each study step.

Protocol: Once enrolled, the patients are ventilated in PS (PScli1) as set by the clinician. They are then ventilated in NAVA at 3 different levels of muscle unloading in randomized order. At NAVAcli, the assist level matches to PScli1 in terms of muscle unloading. With NAVA40% and NAVA60%, the patients have 40% and 60% unloading, respectively. In the last study step the patients are back to PS (PScli2). Each patient is his/her own control and goes through the 5 ventilation periods, of 30min each. In the last 5 min of each study step, the CoV (obtained through the EIT data), blood gas samples (for oxygenation and ventilation) and ventilatory parameters are obtained and analyzed.

The investigators hypothesize that

1. It is possible to set NAVA at different levels of unloading, based on NVE.
2. Moderate muscle unloading (corresponding to NAVA40%) keeps the diaphragm active and thereby leads to more dorsal distribution of ventilation compared to PScli and to higher unloading in NAVA.
3. Secondarily and as a consequence of the redistribution of ventilation, we hypothesize that the gas exchange will remain unchanged or will improve and that the airway pressures will decrease for moderate unloading (NAVA40%).

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to Neurosurgical ICU
* Intubated for ≥48h
* Weaning phase from Mechanical Ventilation

Exclusion Criteria:

* bleeding disorders (PK INR>1,5 or APTT>50s or platelet count <50000/µL) or
* unstable intracranial pressure (ICP>20 mmHg during the latest 8 hours) or
* unstable circulation (requiring high vasopressor dose, for example Noradrenalin >0,2µg/kg/min) or
* too severe lung disease (PFI ≤ 26,7 kPa or PEEP >10 cmH2O or FiO2>0,5 at study entry point) or
* fever> 38,5°C or
* tendency to hyperventilation (PaCO2 < 4,5 kPa at study entry point).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Center of Ventilation (CoV), expressed in percent (ventral to dorsal) | Total study time is 2,5 hours
  The distribution of ventilation is summarized by the CoV, a parameter obtained by the EIT monitor. Recordings are made at the end of each study step (total 5), lasting 30min.

SECONDARY OUTCOMES:
Gas Exchange (PaO2 and PaCO2) | During the last 5min of each study step (each 30min), total 5 steps. Total study time 2,5 hours
  Comparison between study steps
Airway Pressure | 2,5 hours
Muscle unloading based on Neuro-Ventilatory Efficiency and Neuro-Mechanica Efficiency | 2,5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Sackey, MD, PhD, Study Chair — Karolinska University Hospital; Francesca Campoccia Jalde, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Dept. Anesthesiology, Surgical Services and Intensive Care Medicine,Karolinska Univeristy Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Background] Blankman P, Hasan D, van Mourik MS, Gommers D. Ventilation distribution measured with EIT at varying levels of pressure support and Neurally Adjusted Ventilatory Assist in patients with ALI. Intensive Care Med. 2013 Jun;39(6):1057-62. doi: 10.1007/s00134-013-2898-8. Epub 2013 Apr 4. PMID 23553568
- [Background] Liu L, Liu H, Yang Y, Huang Y, Liu S, Beck J, Slutsky AS, Sinderby C, Qiu H. Neuroventilatory efficiency and extubation readiness in critically ill patients. Crit Care. 2012 Jul 31;16(4):R143. doi: 10.1186/cc11451. PMID 22849707
- [Background] Grasselli G, Beck J, Mirabella L, Pesenti A, Slutsky AS, Sinderby C. Assessment of patient-ventilator breath contribution during neurally adjusted ventilatory assist. Intensive Care Med. 2012 Jul;38(7):1224-32. doi: 10.1007/s00134-012-2588-y. Epub 2012 May 15. PMID 22584798
- [Background] Liu L, Liu S, Xie J, Yang Y, Slutsky AS, Beck J, Sinderby C, Qiu H. Assessment of patient-ventilator breath contribution during neurally adjusted ventilatory assist in patients with acute respiratory failure. Crit Care. 2015 Feb 18;19(1):43. doi: 10.1186/s13054-015-0775-2. PMID 25882607